CLINICAL TRIAL: NCT05015257
Title: The Underlying Causes Affecting the Response to Dietary Rehabilitation in Severely Acutely Malnourished Children at the Center Hôspitalier Universitaire Sourô Sanou, Bobo Dioulasso, Burkina Faso
Brief Title: Effectiveness of Four Transition Dietary Regimens in the Hospital Management of Children With Kwashiorkor.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); University Hospital Sourô Sanou of Bobo Dioulasso (Burkina Faso) (Unknown); Centre Muraz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC-09443-B
Record Dates: First submitted 2021-08-02; First posted 2021-08-20 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Severe Acute Malnutrition; Kwashiorkor; Nutritional Edema
Keywords: Severe acute malnutrition; Nutritional rehabilitation; F100; Transition phase; Therapeutic complex of vitamins and minerals (CMV); Kwashiorkor; Ready-to-use Therapeutic Food
MeSH Terms: conditions — Severe Acute Malnutrition; Kwashiorkor

STUDY DESIGN:
Intervention Model Description: This is an open label randomized controlled trial to test the effectiveness of four diets in Kwashiorkor children in their transition phase.
  When it is decided to move to the transition phase, the child will be assigned to one of the treatments depending on the treatment received during the stabilization phase and the results of the appetite test. That is a child who accepts the Plumpy Nut will receive it in combination with their regimen they had during the stabilization phase. If a child does not accept Plumpy Nut, then they will received F100 regardless of their initial therapeutic food regimen.
  * For those who received F75 in the stabilization phase, they will receive standard F75 + Plumpy Nut
  * For those who received alternative F75 with CMV in the stabilization phase, they will receive alternative F75 with CMV + Plumpy Nut®
  * For those who received alternative F75 without CMV in the stabilization phase, they will receive alternative F75 without CMV + Plumpy Nut®.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard F100 (Active Comparator): If the test of appetite at the end of the stabilization phase is negative (the child does not accept the Plumpynut)
  Interventions: Dietary Supplement: Standard F100
- Standard F75+Plumpynut (Experimental): If the test of appetite at the end of the stabilization phase is positive (the child accepts the Plumpynut) and the child received Standard F75 during the stabilization phase
  Interventions: Dietary Supplement: Standard F75 + Plumpynut
- Alternative F75 with CMV +Plumpynut (Experimental): If the test of appetite at the end of the stabilization phase is positive (the child accepts the Plumpynut) and the child received Alternative F75 with CMV during the stabilization phase
  Interventions: Dietary Supplement: Alternative F75 with CMV + Plumpynut
- Alternative F75 without CMV +Plumpynut (Experimental): If the test of appetite at the end of the stabilization phase is positive (the child accepts the Plumpynut) and the child received Alternative F75 without CMV during the stabilization phase
  Interventions: Dietary Supplement: Alternative F75 without CMV + Plumpynut

INTERVENTIONS:
Dietary Supplement: Standard F100 — 100 kcal and 3 g protein per 100 ml
  Arms: Standard F100
Dietary Supplement: Standard F75 + Plumpynut — Standard F75 with ready to-use therapeutic food (Plumpynut)
  Arms: Standard F75+Plumpynut
Dietary Supplement: Alternative F75 with CMV + Plumpynut — Alternative F75 containing CMV with ready to-use therapeutic food (Plumpynut)
  Arms: Alternative F75 with CMV +Plumpynut
Dietary Supplement: Alternative F75 without CMV + Plumpynut — Alternative F75 with no CMV with ready to-use therapeutic food (Plumpynut)
  Arms: Alternative F75 without CMV +Plumpynut

SUMMARY:
In Burkina Faso the number of severely acute malnourished (SAM) children successfully treated has increased since the implementation of community-based management of acute malnutrition. SAM children with oedema have a higher risk of dying than SAM without oedema; they require inpatient care. Several theories have been proposed to explain the pathophysiology of oedema in SAM, but its etiology remains unclear. Knowledge on the nutritional adequacy of therapeutic regimens in kwashiorkor is limited. The World Health Organization (WHO) recommends to use in the treatment of complicated SAM a therapeutic milk 'F75' in the stabilization phase; F75+ready-to-use therapeutic foods (RUTF) or F100 at the transition phase. Alternatively the local formulas (maize flour, milk powder, oil, sugar, mineral-vitamin complex CMV) can be used in case of shortage or intolerance.

At the Nutritional Rehabilitation and Education Center of the University Hospital of Bobo Dioulasso it was found that some SAM children whose oedema resolved under F75 in the stabilization phase, re-developed oedema as they entered the transition phase with RUTF. RUTF has the same nutritional value as F100 but contains iron unlike F100 (<0.07 mg/100 mL). It was observed that RUTF in some cases may be associated with higher mortality, probably due to high iron content (10-14 mg/100 g), which may increase the risk of infections and the formation of free radicals, thereby increasing damage to the body's cells. Clinical trials evaluating the current guidelines for the treatment of SAM with oedema are scarce. A better understanding of the risk factors affecting the effectiveness of the nutritional therapeutic protocol for children with Kwashiorkor will be useful to improve their care.

The main objective of this study is to determine whether the use of transition phase diets (Plumpy-Nut®+F75 or F100 or alternative F75+/- CMV+ Plumpy-Nut®) affect oedema resolving in Kwashiorkor children and to investigate the underlying factors for the relapse or non-responsiveness to the therapeutic treatment.

DETAILED DESCRIPTION:
Severe acute malnutrition (SAM) is a life threatening condition that requires urgent attention and appropriate management to reduce mortality and promote recovery among children. SAM is defined by 1) a weight-for-height Z-score more than three standard deviations (SD) below the median based on the 2006 WHO growth standards, 2) a mid-upper arm circumference (MUAC) of less than 115 mm or 3) by the presence of nutritional edema. Signs such as edema, mucocutaneous changes, hepatomegaly, lethargy, anorexia, anemia, severe immune deficiency and rapid progression to mortality characterize a state commonly coined as "complicated SAM". Kwashiorkor (SAM with edema) is one of the forms of complicated SAM commonly distinguished by the unmistakable presence of bipedal edema. Kwashiorkor is characterized by the following clinical signs: 1) edemas symmetrical, painless, soft, bilateral, ascending, pitting; 2) lesions of the skin and integuments; 3) ulcerations and depigmentation; 4) alopecia; 5) constant weight loss marked by edema; 6) hepatomegaly; 7) clinical anemia; 8) intestinal transit disorders: persistent diarrhea, vomiting; 9) anorexia and behavioral disorders (apathy).

Severe acute malnutrition results in high mortality rates of up to half a million child deaths annually. Undernourished children are at higher risk of mortality ranging from three-times more risk among children with moderate malnutrition to 10-times in SAM children compared to well-nourished children.

The objective of this study is to determine whether the use of different transition phase diets affect oedema resolving in Kwashiorkor children and to investigate the underlying factors for the relapse or non-responsiveness to the therapeutic treatment.

Hypotheses to be tested

* The first hypothesis is that RUTF (Plumpy-Nut®) because of its content in iron may compromise the effectiveness of the transition phase in children with kwashiorkor
* The second hypothesis is that underlying factors including co-morbidities and epigenetics may explain a difference in response to therapeutic regimens

This is an open label randomized controlled trial to test the effectiveness of four used transition phase diets in Kwashiorkor children in their transition to the rehabilitation phase. The four dietary regimens that will be tested are:

1. F100;
2. RUTF+F75;
3. RUTF+alternative F75 with complex mineral-vitamin (CMV); and
4. RUTF+alternative F75 without CMV.

When it is decided to move to the transition phase, the child will be assigned to one of the treatments depending on the treatment received during the stabilization phase and the results of the appetite test. That is a child who accepts the Plumpy Nut will receive it in combination with their regimen they had during the stabilization phase. If a child does not accept Plumpy Nut, then they will received F100 regardless of their initial therapeutic food regimen.

* For those who received F75 in the stabilization phase, they will receive standard F75 + Plumpy Nut
* For those who received alternative F75 with CMV in the stabilization phase, they will receive alternative F75 with CMV + Plumpy Nut®
* For those who received alternative F75 without CMV in the stabilization phase, they will receive alternative F75 without CMV + Plumpy Nut®.

ELIGIBILITY:
Inclusion Criteria:

* Severe acute malnutrition defined as the presence of edema
* Who are admitted and treated in the refeeding center (CREN) of the CHUSS
* Aged between 6 and 59 Months
* Parental Signed informed consent form
* Recruited in the first phase of the treatment and successfully admitted to the transition phase

Exclusion Criteria:

* SAM without edema
* Moderate acute malnutrition (MAM)
* Did not improve during the stabilization phase

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Edema redevelopment during the transition phase | Three to Seven days
  Number of children whose edema redeveloped after it has been resolved during the stabilization phase
Severe adverse event | Three to Seven days
  Any serious severe adverse event ranging from diarrhea, vomiting, anorexia to death

SECONDARY OUTCOMES:
Mean number of days for a complete edema resolving | Three to Seven days
  Number of days for a complete edema resolving among Kwashiorkor children, in Day
Intestinal microbiota | Three to Seven days
  16S rRNA sequencing of DNA extracts of fecal samples
Presence of acidic stools | Three to Seven days
  Measurement of stool potential Hydrogen (pH)
Soil Helminths | Three to Seven days
  Determination of intestinal parasites using Quantitative Real-Time polymerase chain reaction (qPCR)
Epigenetics | Three to Seven days
  In a subsample of children, DNA methylation is identified using Illumina Array Analysis Platform

CONTACTS AND LOCATIONS:
Overall Officials: Stefaan De Henauw, Md. PhD, Principal Investigator — University Ghent; Souheila Abbeddou, MSc. PhD, Principal Investigator — University Ghent; Jerome Some, Md. PhD, Principal Investigator — Institut de Recherche en Sciences de la Sante, Burkina Faso; Bintou Sanogo, MSc. Md., Principal Investigator — Centre Hospitalier Universitaire Souro, Bobo Dioulasso, Burkina Faso.
Locations (1):
- Centre Hospitalier Universitaire Souro, Bobo-Dioulasso, Bobo Dioulasso, Burkina Faso

IPD SHARING:
Plan to Share IPD: No
All the data that can affect the main or the secondary outcomes will be used in the analyses and shared as necessary

REFERENCES:
- [Background] Gopalan C. Kwashiorkor and marasmus: evolution and distinguishing features. 1968. Natl Med J India. 1992 May-Jun;5(3):145-51. No abstract available. PMID 1306670
- [Background] Nguefack F, Adjahoung CA, Keugoung B, Kamgaing N, Dongmo R. [Hospital management of severe acute malnutrition in children with F-75 and F-100 alternative local preparations: results and challenges]. Pan Afr Med J. 2015 Aug 31;21:329. doi: 10.11604/pamj.2015.21.329.6632. eCollection 2015. French. PMID 26587175
- [Background] Singh K, Badgaiyan N, Ranjan A, Dixit HO, Kaushik A, Kushwaha KP, Aguayo VM. Management of children with severe acute malnutrition: experience of Nutrition Rehabilitation Centers in Uttar Pradesh, India. Indian Pediatr. 2014 Jan;51(1):21-5. doi: 10.1007/s13312-014-0328-9. Epub 2013 Jul 5. PMID 24277964
- [Background] Smith MI, Yatsunenko T, Manary MJ, Trehan I, Mkakosya R, Cheng J, Kau AL, Rich SS, Concannon P, Mychaleckyj JC, Liu J, Houpt E, Li JV, Holmes E, Nicholson J, Knights D, Ursell LK, Knight R, Gordon JI. Gut microbiomes of Malawian twin pairs discordant for kwashiorkor. Science. 2013 Feb 1;339(6119):548-54. doi: 10.1126/science.1229000. Epub 2013 Jan 30. PMID 23363771
- See also: World Health Organization (2013) WHO guideline: updates on the management of severe acute malnutrition in infants and children — https://www.who.int/publications/i/item/9789241506328
- See also: Enquête Nutritionnelle Nationale SMART 2016 au Burkina Faso. 2016 ; 47p — https://www.unicef.fr/article/malnutrition-la-situation-au-burkina-faso
- See also: Ministère de la Sante au Burkina Faso. Protocol National : Prise en charge intégrée de la malnutrition aigüe (PCIMA). 2014 — https://www.humanitarianresponse.info/sites/www.humanitarianresponse.info/files/documents/files/protocole_pcima_bf_janv_2015.pdf